CLINICAL TRIAL: NCT02558322
Title: Regional Variation of Patient Population and Reasons for Consultation in the Primary Medical Care of Northern Germany
Brief Title: Regional Variation in the Primary Medical Care of Northern Germany
Acronym: AVFN
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: KVHH-KVSH-2015/1
Record Dates: First submitted 2015-09-02; First posted 2015-09-24 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Any Condition Treated in Primary Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Primary medical care in rural areas: People living in districts, where less than 50% of the population live in cities with more than 20,000 residents and the population density outside of the cities is below 100 people per km². Excluding people living in cities with a population of at least 100,000 residents.
  Interventions: Other: Primary medical care
- Primary medical care in region environs: People living in districts, where 50% or more of the population live in cities with more than 20,000 residents and/or population density outside of the cities is above 100 people per km². Excluding people living in cities with a population of at least 100,000 residents.
  Interventions: Other: Primary medical care
- Primary medical care in in urban areas: People living in cities with a population of at least 100,000 residents.
  Interventions: Other: Primary medical care

INTERVENTIONS:
Other: Primary medical care — All study participants receive primary care as usual in the respective region

SUMMARY:
The study explores the variation in the patient populations and describes regional differences regarding the reasons for consultations in the primary medical care in Germany. The data collection will be stratified by rural and urban areas as well as environs. The data set will include a large variety of data about physicians, patients and health care utilization.

DETAILED DESCRIPTION:
Inappropriate supply and the increasing demand on the health care system have been of concern for health policy in Germany for the last 15 years. Concerning primary care, this especially relates to an undersupply of rural GPs (general practitioners). But there also seem to be other relevant regional differences, e.g. a lower number of house calls in larger cities, a greater number of psychiatric (co-)morbidities in the cities, a greater spectrum of services offered by rural doctors, and a difference in accessing primary and secondary care between the rural and the urban areas. Despite these results, differences between rural and urban areas have not been studied extensively in Germany. Therefore this study aims to explore regional variation of patient populations and their reasons for accessing primary care.

The study is based on standardized interviews with 240 GPs and approximately 1.200 patients in Northern Germany. Questionnaires are based on a preliminary qualitative study and were pretested. The GP's questionnaire comprises characteristics of the GP and the practice, patient types, reasons for consultation and services offered. The patient's questionnaire includes sociodemographic data and past medical history, quality of life, access to the GP, specialists and hospitals, perceived social support, health behaviour and the reasons for their consultations. Data will be analysed by descriptive statistics and different regression modelling strategies adjusted for possible confounders and the GP-induced cluster structure.

ELIGIBILITY:
Inclusion Criteria:

* having consulted the practice within the last 3 months and
* being patient of the practice since at least 36 months (i.e. at least one consultation before 36 or more months)

Exclusion Criteria:

* no capacity to consent (e.g. because of dementia)
* insufficient German language skills to conduct interview
* not able to participate in the interviews (e.g. because of deafness or major depression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is located in Northern Germany. We included all districts and cities ("Landkreise" and "Kreisfreie Städte") which have at least 20% of their area within a maximum linear distance of 100kms from our study centre in Hamburg. We assigned all districts and cities to three region types: "urban area", "environs" and "rural area". In each region type 80 GPs will be recruited and stratified by district. The prospected sample size in each district unit corresponds to its population size in relation to the total population in the respective region type. In each GP practice 15 patients will be selected at random (using random number tables) and invited to participate in the study. From our experience with similar studies we anticipate a response rate of 33%.
Sampling Method: Probability Sample
Enrollment: 1022 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Reasons for consultation and utilized services in the GP practice | 3 months
  Short form of the German version of the International Classification of Primary Care (ICPC) with 38 different services (e.g. vaccinations, patient education or referrals) and 100 consultation reasons (e.g. disorders of the upper gastrointestinal tract) in 17 subject areas (e.g. digestive system).

SECONDARY OUTCOMES:
Patient population in the GP practice | 3 months
  List of 27 patient types regarding their health care utilization behaviour
Health care utilization | 3 months
  Frequency of accessing GPs, specialists, general hospitals and rehab hospitals

CONTACTS AND LOCATIONS:
Overall Officials: Martin Scherer, Prof. Dr., Principal Investigator — Department of Primary Medical Care, University Medical Center Hamburg-Eppendorf
Locations (1):
- Department of Primary Medical Care, University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Derived] Hansen H, Schafer I, Pohontsch NJ, Kazek A, Hardt H, Luhmann D, Scherer M. Regional differences in the patient population of general practices in northern Germany: results of a mixed-methods study. BMJ Open. 2020 Nov 27;10(11):e041762. doi: 10.1136/bmjopen-2020-041762. PMID 33247029
- [Derived] Hansen H, Schafer I, Porzelt S, Kazek A, Luhmann D, Scherer M. Regional and patient-related factors influencing the willingness to use general practitioners as coordinators of the treatment in northern Germany - results of a cross-sectional observational study. BMC Fam Pract. 2020 Jun 17;21(1):110. doi: 10.1186/s12875-020-01180-3. PMID 32552721
- [Derived] Schafer I, Hansen H, Ruppel T, Luhmann D, Wagner HO, Kazek A, Scherer M. Regional differences in reasons for consultation and general practitioners' spectrum of services in northern Germany - results of a cross-sectional observational study. BMC Fam Pract. 2020 Jan 31;21(1):22. doi: 10.1186/s12875-020-1093-6. PMID 32005159
- [Derived] Schafer I, Hansen H, Pohontsch N, Bole L, Wagner HO, Fuhr M, Luhmann D, Scherer M. Regional variation of patient behaviour and reasons for consultation in the general practice of Northern Germany: protocol for an observational study. BMJ Open. 2016 Jun 29;6(6):e010738. doi: 10.1136/bmjopen-2015-010738. PMID 27357194